CLINICAL TRIAL: NCT05510089
Title: Prospective, Single-arm, Multicenter Exploratory Clinical Study of the Combination of Etoposide, Cytarabine and PEG-rhG-CSF (EAP Regimen) on Hematopoietic Stem Cell Mobilization in Poor Mobilization Patients With Hematological Malignancies
Brief Title: Etoposide+Cytarabine+PEG-rhG-CSF for Hematopoietic Stem Cell Mobilization in Patients With Hematological Malignancies
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: The Affiliated People's Hospital of Ningbo University (Other Government)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2022-YAN-019
Record Dates: First submitted 2022-08-18; First posted 2022-08-22 (Actual); Last update posted 2023-10-10 (Actual); Status verified 2023-08

CONDITIONS: Hematological Malignancy
Keywords: Etoposide; Cytarabine; PEG-rhG-CSF; Hematological Malignancies; Hematopoietic Stem Cell Mobilization
MeSH Terms: conditions — Hematologic Neoplasms | interventions — Etoposide; Cytarabine; pegylated granulocyte colony-stimulating factor

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- EAP regimen (Experimental): The combination regimen of etoposide, cytarabine and PEG-rhG-CSF.
  Interventions: Drug: Etoposide; Drug: Cytarabine; Drug: PEG-rhG-CSF

INTERVENTIONS:
Drug: Etoposide — D1~D2: 75mg/m^2
  Other Names: VP-16
Drug: Cytarabine — D1~D2: 300mg/m^2, q12h
  Other Names: Ara-C
Drug: PEG-rhG-CSF — D6: 6mg

SUMMARY:
This is a single-arm, multicenter, exploratory clinical study to evaluate the safety and efficacy of the combination of etoposide, cytarabine and PEG-rhG-CSF (EAP regimen) on hematopoietic stem cell mobilization in poor mobilization patients with hematological malignancies. All eligible patients will receive EAP regimen treatment, then the number of CD34+ cells and white blood cells will be monitoring. When the collection standard is met, hematopoietic stem cell collection will be started.

ELIGIBILITY:
Inclusion Criteria:

1. According to the diagnostic criteria of the Italian transplantation working group, patients with multiple myeloma or lymphoma diagnosed as "confirmed poor mobilization" or "predicted poor mobilization".
2. Patients with auto-HSCT indication.
3. Eastern Cooperative Oncology Group (ECOG) performance status of 0~2.
4. Patients should be within age range of ≥18 and ≤75 years old.
5. Life expectancy ≥ 3 months.
6. Patients must be able to sign informed consent.

Exclusion Criteria:

1. Patients with severe cardiac, hepatic or renal insufficiency, such as:

   * Cardiac function class II or higher or severe arrhythmia;
   * Serum direct bilirubin (DBIL)>2× upper limit of normal (ULN);
   * Aspartate aminotransferase (AST) or alanine aminotransferase (ALT) > 2× ULN;
   * Serum creatinine clearance rate≤50%.
2. Patients with active infection.
3. History of allergy to Etoposide (VP-16), Cytarabine (Ara-C), or PEG-rhG-CSF.
4. Women who are pregnant or breastfeeding.
5. Have received live vaccine and attenuated live vaccine within 4 weeks before enrollment.
6. For any other reasons, the patients are believed not suitable for participation in this study by investigators

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 62 (Estimated)
Dates: Start 2022-09-01 (Actual); Primary Completion 2024-05-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
% of patients achieving the collection of ≥2×10^6 CD34+ cells/kg. | 4 weeks
  The proportion of patients whose cells can be successfully mobilized and collected with a target CD34+ Hematopoietic Stem Cell (HSC) dose of ≥2×10^6/kg.

SECONDARY OUTCOMES:
% of patients achieving the collection of >5×10^6 CD34+ cells/kg. | 4 weeks
  The proportion of patients whose cells can be successfully mobilized and collected with a target CD34+ Hematopoietic Stem Cell (HSC) dose of >5×10^6/kg.
TRAEs | 4 weeks
  Incidence and severity of treatment related adverse events (TRAEs). Adverse events will be collected based on NCI CTCAE version 5.0.
Time from PEG-rhG-CSF mobilization to HSC collection. | 4 weeks
  To determine the time period from PEG-rhG-CSF mobilization to successfully collection of HSC.
The average collection times of EAP regimen | 4 weeks
Hematopoietic reconstitution and therapeutic adverse events after transplantation | 4 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Ying Lu, Principal Investigator — The Affiliated People's Hospital of Ningbo University
Locations (12):
- China (12):
  - Dongyang People's Hospital, Dongyang, Zhejiang
  - Tongde Hospital of Zhejiang Province, Hangzhou, Zhejiang
  - The First Affiliated Hospital, Zhejiang University School of Medicine, Hangzhou, Zhejiang
  - Huzhou central hospital, Huzhou, Zhejiang
  - Jinhua Municipal Central Hospital, Jinhua, Zhejiang
  - Jinhua People's Hospital, Jinhua, Zhejiang
  - Lishui Municipal Central Hospital, Lishui, Zhejiang
  - The Affiliated People's Hospital of Ningbo University., Ningbo, Zhejiang
  - Shaoxing People's Hospital, Shaoxing Hospital of Zhejiang University, Shaoxing, Zhejiang
  - Shaoxing Second Hospital, Shaoxing, Zhejiang
  - Taizhou Central Hospital, Taizhou, Zhejiang
  - Taizhou Hospital of Zhejiang Province, Taizhou, Zhejiang